CLINICAL TRIAL: NCT04626869
Title: Anterior Suprascapular Nerve Block is as Effective as Interscalene Nerve Block and Causes Less Diapragm Paralysis in Arthroscopic Shoulder Surgery
Brief Title: Anterior Suprascapular Nerve Block is an Effective and Diaphragm Protective Approach for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alper Tunga Dogan (Other)
Responsible Party: Sponsor-Investigator, Alper Tunga Dogan, Anesthesiology specialist, V.K.V. American Hospital, Istanbul
Organization: V.K.V. American Hospital, Istanbul (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.1234
Record Dates: First submitted 2020-09-16; First posted 2020-11-13 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Diaphragm Paralysis Due to Local Anesthesia; Anterior Suprascapular Nerve Block; Analgesia, Arthroscopic Shoulder Surgery
Keywords: arthroscopic shoulder surgery; Interscalene nerve block; Anterior suprascapular nerve block; Analgesia, postoperative; Diaphragm paralysis
MeSH Terms: conditions — Agnosia; Respiratory Paralysis

STUDY DESIGN:
Intervention Model Description: The patients will be divided into two groups as patients who underwent suprascapular nerve block with the supraclavicular approach and patients who underwent conventional interscalene nerve block. 5 ml of 0.5% Bupivacaine will be injected into both groups. Diaphragmatic movement will be evaluated with ultrasound at the right and left subcostal border with the patients in a semi-sitting position. The reduction in diaphragm motion will be calculated as the difference (in percent) in diaphragm motion measured before and 30 minutes after the block.
Who Masked: Outcomes Assessor
Masking Description: Diaphragm Measurements will be done by an expert unaware of the working groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block (Active Comparator): patients will be placed in a semi-sitting position with their heads facing the opposite side. Linear ultrasound probe (GE Loqic P9 7-15 MHz) to detect the brachial plexus. At the cervical level 5-6, the posterior brachial plexus will be approached as "in-plane" from the posterior with the needle (Contiplex C, Braun) through the catheter. The nerve structure will be confirmed with stimulation in the upper extremity muscles with a nerve stimulator and 5 ml 0.5% Bupivacaine will be injected.
  Interventions: Other: Evaluation of Diaphragm Movement
- Anterior suprascapular nerve block (Active Comparator): patients will be placed in a semi-sitting position with their heads facing the opposite side. Linear ultrasound probe (GE Loqic P9 7-15 MHz) will be placed in the suprascapular region in a coronal oblique manner. The omohyoid muscle, under it the suprascapular nerve, the brachial plexus and the subclavian artery will be identified. The suprascapular nerve will be approached from the posterior as "in-plane" with a needle (Contiplex C, Braun) through the catheter. The nerve structure will be confirmed by stimulation in the supraspinous muscle with a nerve stimulator and 5 ml 0.5% Bupivacaine will be injected.
  Interventions: Other: Evaluation of Diaphragm Movement

INTERVENTIONS:
Other: Evaluation of Diaphragm Movement — Diaphragmatic movement will be evaluated with ultrasonography and a 5-2 MHz convex transducer will be used. The ultrasound probe is placed between the mid-clavicular line and the anterior axillary line by directing it vertically and slightly cranially. During quiet breathing and deep breathing, diaphragm movement will be measured. The reduction in diaphragm motion will be calculated as the difference (in percent) in diaphragm motion measured before and 30 minutes after the block. Each test will be done 3 times and the values will be averaged. A decrease between 75% and 100% will be defined as complete paresis, a decrease between 25% and 75% as partial paresis, and less than 25% decrease in diaphragmatic movement will be defined as no paresis. In order to investigate the effect of continuous local anesthetic drug administration on diaphragm movement via nerve catheter, the same procedure will be repeated 24 hours after surgery.

SUMMARY:
Interscalene block is still the gold standard in shoulder surgery analgesia. The most important side effect is diaphragm paralysis due to the phrenic nerve being affected. It may cause symptomatic dyspnea, especially in patients with limited respiratory capacity. There are studies showing that an effective analgesia, as much as the interscalene block can do, can be provided by blocking the suprascapular nerve in the neck region.

The aim of our study is to show that the anterior suprascapular block applied with ultra-low volume (5ml) in shoulder arthroscopy operations is at least as effective as the interscalene block and does not cause diaphragm paralysis.

DETAILED DESCRIPTION:
Interscalene block is still the gold standard in shoulder surgery analgesia. The most important side effect is diaphragm paralysis due to the phrenic nerve being affected. It may cause symptomatic dyspnea, especially in patients with limited respiratory capacity. More distal brachial plexus blocks have been defined to avoid diaphragmatic paralysis . Thus, it is aimed to apply the local anesthetic drug further from the phrenic nerve. With the application of ultrasound, the amount of local anesthetic drug was reduced to less than 20 ml.

There are studies showing that an effective analgesia, as much as the interscalene block can do, can be provided by blocking the suprascapular nerve in the neck region. Although it has been shown in a cadaver study that the phrenic nerve can be stained after anterior suprascapular nerve block, the clinical effect is not fully known.

The effect of continuous local anesthetic drug administration on respiratory muscles through catheters placed in the peripheral nerve is another matter of concern. The method that will not affect the phrenic nerve at all and at the same time provide an effective analgesia is still under investigation.

The aim of our study is to show that the anterior suprascapular block applied with ultra-low volume (5ml) in shoulder arthroscopy operations is at least as effective as the interscalene block and does not cause diaphragm paralysis. One of the questions that our research aims to answer is how the continuous application of local anesthetic drugs affects the diaphragm muscle with the insertion of catheters in both regions.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* American Society of Anesthesiology (ASA) score of 1-3
* Scheduled for elective surgery.

Exclusion Criteria:

* Patients with a condition that prevents peripheral nerve block
* Coagulopathies
* Chronic opioid use
* Stroke
* Polyneuropathy
* Cognitive dysfunction
* Communication difficulties
* Allergies to drugs used

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Pain rating | the first postoperative 30 minutes
  Measured by VAS. Postoperative 30 minutes
Pain rating | Postoperative 6 hours
  Measured by VAS. Postoperative 6 hours
Pain rating | Postoperative 12 hours
  Measured by VAS. Postoperative 12 hours

SECONDARY OUTCOMES:
Diaphragmatic movements | 30 minutes after the block application.
  Diaphragmatic movement will be evaluated with ultrasound. 30 minutes after the block application.
Diaphragmatic movements | At the first postoperative 24 hours
  Diaphragmatic movement will be evaluated with ultrasound. 24 hours after the block application.

CONTACTS AND LOCATIONS:
Locations (1):
- VKV Amerikan Hastanesi, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tran DQ, Layera S, Bravo D, Cristi-Sanchez I, Bermudez L, Aliste J. Diaphragm-sparing nerve blocks for shoulder surgery, revisited. Reg Anesth Pain Med. 2019 Sep 20:rapm-2019-100908. doi: 10.1136/rapm-2019-100908. Online ahead of print. PMID 31541010
- [Result] Bansal V, Shastri U, Canlas C, Gadsden JC. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery: An Alternative Approach. Reg Anesth Pain Med. 2017 Jul/Aug;42(4):544-545. doi: 10.1097/AAP.0000000000000606. No abstract available. PMID 28632682
- [Result] Auyong DB, Hanson NA, Joseph RS, Schmidt BE, Slee AE, Yuan SC. Comparison of Anterior Suprascapular, Supraclavicular, and Interscalene Nerve Block Approaches for Major Outpatient Arthroscopic Shoulder Surgery: A Randomized, Double-blind, Noninferiority Trial. Anesthesiology. 2018 Jul;129(1):47-57. doi: 10.1097/ALN.0000000000002208. PMID 29634491
- [Result] Wiegel M, Moriggl B, Schwarzkopf P, Petroff D, Reske AW. Anterior Suprascapular Nerve Block Versus Interscalene Brachial Plexus Block for Shoulder Surgery in the Outpatient Setting: A Randomized Controlled Patient- and Assessor-Blinded Trial. Reg Anesth Pain Med. 2017 May/Jun;42(3):310-318. doi: 10.1097/AAP.0000000000000573. PMID 28257388